CLINICAL TRIAL: NCT03427346
Title: Prospektiv-randomisierter Vergleich Von En-bloc- Versus Piecemeal-Resektion Von Barrett Neoplasien Des Ösophagus Neoplastic Barrett Esophagus: Endoscopic Piecemeal vs. En Bloc Resection
Brief Title: Neoplastic Barrett Esophagus: Endoscopic Piecemeal vs. En Bloc Resection
Acronym: BEEPER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Director of Department of Interdisciplinary Endoscopy, University Medical Center Hamburg-Eppendorf, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PV5387
Record Dates: First submitted 2017-11-08; First posted 2018-02-09 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Barrett Esophagus; Barrett Adenocarcinoma; Esophagus Neoplasm
Keywords: Barrett Esophagus; ESD; EMR; Esophagus Neoplasm; endoscopic resection technique; ablation of esophageal mucosa
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMR (Active Comparator): Endoscopic mucosal resection
  Interventions: Procedure: Endoscopic mucosal resection
- ESD (Active Comparator): Endoscopic submucosal dissection
  Interventions: Procedure: Endoscopic submucosal dissection

INTERVENTIONS:
Procedure: Endoscopic mucosal resection — Endoscopic resection is carried out using a double-channel scope. The lesion borders are marked with a coagulator. Saline liquid and sometimes epinephrine are injected into the submucosal layer to swell the area containing the lesion and elucidate the markings. The resected mucosa is lifted, then trapped and strangulated with a snare, and subsequently resected by electrocautery. Another method of EMR employs the use of a clear cap and prelooped snare inside the cap. After insertion, the cap is placed on the lesion and the mucosa containing the lesion is drawn up inside the cap by aspiration. The mucosa is caught by the snare and strangulated, and finally resected by electrocautery.
  Other Names: EMR; Piecemeal EMR
  Arms: EMR
Procedure: Endoscopic submucosal dissection — After circumferential cutting of the surrounding mucosa of the lesion, fluid is injected into the submucosa to elevate the lesion from the muscle layer, and the connective tissue of the submucosa beneath the lesion is dissected subsequently.
  Other Names: ESD
  Arms: ESD

SUMMARY:
The study will compare EMR versus ESD technique (both combined with subsequent ablative therapy) of mucosal resection in Barrett's esophagus with regard to efficacy and risk in a long term setting.

DETAILED DESCRIPTION:
For Barrett's Esophagus neoplasia of at least LGIN up to early adenocarcinoma, the aim is to debulk or completely treat polypoid dysplastic or malignant lesions in Barrett's esophagus. The Endoscopic Mucosal Resection EMR has been established to be a less invasive, safe, and effective nonsurgical therapy. The most commonly employed modalities of EMR include snare resection with and without prior submucosal injection of fluid, and resection using a cap. Since resection of larger areas can only be done piece - by- piece this kind or resection is also called piecemeal resection or piecemeal EMR. Meanwhile, another endoscopic resection has been developed called Endoscopic Submucosal Dissection ESD.It enables complete resection of neoplasms that were impossible to resect en bloc by EMR. After circumferential cutting of the surrounding mucosa of the lesion, fluid is injected into the submucosa to elevate the lesion from the muscle layer, and subsequently the connective tissue beneath the lesion is dissected. As a basic principle on histopathological and oncological terms, the en bloc resection is to be preferred since resection integrity can be evaluated much more securely. However, complexity of this kind of resection technique as well as complication rates can be different and sometimes higher than with EMR. Current approach treating Barrett's esophagus is to eradicate both neoplastic as well as pre neoplastic or non neoplastic Barrett mucosa in order to lower the relapse risk. Current treatment standard is to combine resection of visible neoplastic areas with subsequent thermo-ablation such as RFA or APC, so this approach will also be the basis of the present study. Since RFA has the largest volume of data screened it shall be the preferred method of ablation in this study.In total, data situation ist inconsistent. Short- and Long term of EMR is excellent in centres(Pech et al, Gastroenterology 2014) whereas ESD achieved only suboptimal outcomes in tree minor western studies (Neuhaus et al. Endoscopy 2012, Höbel et al., Surg Endosc 2015, Chevaux et al. Endoscopy 2015). One randomised study published in 2016 (Terheggen et al. Gut 2016) had a higher rate of R0 resections with ESD on 40 patients but no difference in complete remissions in combination with RFA. Although, this study was not empowered sufficientliy, and also showed a higher complication rate on ESD . At present no randomised study data are availale to allow statements about long term developments, so we will set up this current randomised study. We will compare data with regard to efficacy (histological completeness and relapse rates), as well as risks, e.g. perforations and strictures or stenosis by scarring.

ELIGIBILITY:
Inclusion Criteria:

* patients to be treated for Barrett's esophagus by mucosal resection and following ablative therapy
* Barrett's mucosal extension up to 10 cm maximum.
* patient's ability for compliance to therapy
* signed Informed Consent

Exclusion Criteria:

* any lesion questionable to be resectable by mucosectomy, e.g. bulky lesions ≥10 mm in endoscopy und endosonography, suspected deep submucosal infiltration, ulcers, suspected or by FNA confirmed lymph node infiltration
* Barrett's esophagus > 10 cm
* lesions that would afford resection of more than 2/3rd of esophagal circumference
* two or more single Barrett's lesions with bulky HGIN or early cancer histology, not to be resectable in one half of esophageal circumference
* planned circumferencial resections
* very serious general illness and metastatic carcinoma
* coagulation disorder or anticoagulants that make biopsies and resections impossible
* American Society of Anesthesiologists (ASA) status > III
* pregnancy and lactation
* remainders or recurrences after therapeutic history of Barrett's espohagus

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of neoplastic Barrett's Esophagus, initial therapy success | 3 months after end of therapy (resection and ablation)
  Rate of complete and curative eradication, free of recurrence of neoplastic Barrett's Esophagus. Endoscopical diagnostic and negative histologies for any kind of neoplasia, measured in follow up control EGD 3 months after end of treatment
Eradication rate of neoplastic Barrett's Esophagus, initial therapy success | 9 months after end of therapy (resection and ablation)
  Rate of complete and curative eradication, free of recurrence of neoplastic Barrett's Esophagus. Endoscopical diagnostic and negative histologies for any kind of neoplasia, measured in follow up control EGD 9 months after end of treatment
Eradication rate of neoplastic Barrett's Esophagus | 24 months after end of therapy (resection and ablation)
  Rate of complete and curative eradication, free of recurrence of neoplastic Barrett's Esophagus. Endoscopical diagnostic and negative histologies for any kind of neoplasia, measured in follow up control 24 months after end of treatment
Eradication rate of neoplastic Barrett's Esophagus | 33 months after end of therapy (resection and ablation)
  Rate of complete and curative eradication, free of recurrence of neoplastic Barrett's Esophagus. Endoscopical diagnostic and negative histologies for any kind of neoplasia, measured in follow up control EGD 33 months after end of treatment

SECONDARY OUTCOMES:
Eradication rate of complete Barrett's Esophagus, initial therapy success | 3 months after end of treatment (resection and ablation)
  Rate of complete and curative eradication, free of recurrence of neoplastic and non-neoplastic Barrett's Esophagus. Endoscopical diagnostics and negative histologies for any kind of neoplasia and Barrett's metaplasia measured in follow up control EGD 3 months after end of treatment
Eradication rate of complete Barrett's Esophagus, initial therapy success | 9 months after end of treatment (resection and ablation)
  Rate of complete and curative eradication, free of recurrence of neoplastic and non-neoplastic Barrett's Esophagus. Endoscopical diagnostics and negative histologies for any kind of neoplasia and Barrett's metaplasia measured in follow up control EGD 9 months after end of treatment
Eradication rate of complete Barrett's Esophagus, freedom of recurrence | 24 months after end of treatment (resection and ablation)
  Rate of complete and curative eradication, free of recurrence of neoplastic and non-neoplastic Barrett's Esophagus. Endoscopical diagnostics and negative histologies for any kind of neoplasia and Barrett's metaplasia measured in follow up control EGD 24 months after end of treatment
Eradication rate of complete Barrett's Esophagus, freedom of recurrence | 33 months after end of treatment (resection and ablation)
  Rate of complete and curative eradication, free of recurrence of neoplastic and non-neoplastic Barrett's Esophagus. Endoscopical diagnostics and negative histologies for any kind of neoplasia and Barrett's metaplasia measured in follow up control EGD 33 months after end of treatment
Recurrence rate of neoplastic Barrett's Esophagus, initial therapy success | 3 months after end of therapy (resection and ablation)
  rate of complete and curative eradication of neoplastic Barrett's Esophagus measured in follow up control EGD 3 months, Endoscopical diagnostic and negative histologies for any kind of neoplasia.
Recurrence rate of neoplastic Barrett's Esophagus, initial therapy success | 9 months after end of therapy (resection and ablation)
  rate of complete and curative eradication of neoplastic Barrett's Esophagus measured in follow up control EGD 9 months , Endoscopical diagnostic and negative histologies for any kind of neoplasia.
freedom of recurrence rate of complete Barrett's Esophagus, initial therapy success | 9 months after end of treatment (resection and ablation)
  Freedom of recurrence rate of neoplastic and non-neoplastic Barrett's Esophagus. Endoscopical diagnostics and negative histologies for any kind of neoplasia and Barrett's metaplasia measured in follow up control EGD 9 months (initial therapy success) after end of treatment
ESD success of resection | 2 days
  rate of en bloc and R0 resections among the initially by ESD resected tissues
EMR success of resection | 9 months after end of treatment (resection and ablation)
  Since with EMR resection success can only be measured for the depth of base initially, the second control EGD with negative histology has been chosen for Gold standard indication for resection success. After 2 negative bioptic controls a piecemeal resection of early carcinoma is classified as complete.
Surveillance of Barrett's mucosa after incomplete resections and recurrences | 51 months
  follow up of all cases with initially incomplete EMR or ESD resections as well as recurrences after resection and ablation
conclusions of Tumor Board in case of re resection and outcome if postitive cancer histology | 51 months
  any Treatment and follow up in case of positive cancer histology
Determination of differences in Barrett's esophagus subtypes: size | 3 months
  size of Barrett's mucosa, e.g. Prague Classification
Determination of differences in Barrett's esophagus subtypes: form | 3 months
  form of Barrett's mucosa
Determination of differences in Barrett's esophagus subtypes: patterns | 3 months
  patterns of Barrett's mucosa, e,g, Kudo Classification
Determination of differences in Barrett's esophagus subtypes: histologies | 3 months
  histological assessment of Barrett's mucosa
Intervention time | 18 months
  time requested for each resection and ablative sessions

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, Prof. Dr., Principal Investigator — Ph D, Director, Head of department
Locations (2):
- Orlando Health, Orlando, Florida, United States
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anders M, Bahr C, El-Masry MA, Marx AH, Koch M, Seewald S, Schachschal G, Adler A, Soehendra N, Izbicki J, Neuhaus P, Pohl H, Rosch T. Long-term recurrence of neoplasia and Barrett's epithelium after complete endoscopic resection. Gut. 2014 Oct;63(10):1535-43. doi: 10.1136/gutjnl-2013-305538. Epub 2014 Jan 3. PMID 24389236
- [Background] BARRETT NR. The oesophagus lined by columnar epithelium. Gastroenterologia. 1956;86(3):183-6. doi: 10.1159/000200553. No abstract available. PMID 13384591
- [Background] BARRETT NR. The lower esophagus lined by columnar epithelium. Surgery. 1957 Jun;41(6):881-94. No abstract available. PMID 13442856
- [Background] Dunbar KB, Spechler SJ. Controversies in Barrett esophagus. Mayo Clin Proc. 2014 Jul;89(7):973-84. doi: 10.1016/j.mayocp.2014.01.022. Epub 2014 May 24. PMID 24867396
- [Background] Edgren G, Adami HO, Weiderpass E, Nyren O. A global assessment of the oesophageal adenocarcinoma epidemic. Gut. 2013 Oct;62(10):1406-14. doi: 10.1136/gutjnl-2012-302412. Epub 2012 Aug 23. PMID 22917659
- [Background] Hobel S, Dautel P, Baumbach R, Oldhafer KJ, Stang A, Feyerabend B, Yahagi N, Schrader C, Faiss S. Single center experience of endoscopic submucosal dissection (ESD) in early Barrett's adenocarcinoma. Surg Endosc. 2015 Jun;29(6):1591-7. doi: 10.1007/s00464-014-3847-5. Epub 2014 Oct 8. PMID 25294533
- [Background] Labenz J, Koop H, Tannapfel A, Kiesslich R, Holscher AH. The epidemiology, diagnosis, and treatment of Barrett's carcinoma. Dtsch Arztebl Int. 2015 Mar 27;112(13):224-33; quiz 234. doi: 10.3238/arztebl.2015.0224. PMID 25869347
- [Background] Neuhaus H. Endoscopic mucosal resection and endoscopic submucosal dissection in the West--too many concerns and caveats? Endoscopy. 2010 Oct;42(10):859-61. doi: 10.1055/s-0030-1255724. Epub 2010 Sep 30. No abstract available. PMID 20886404
- [Background] Pech O, May A, Manner H, Behrens A, Pohl J, Weferling M, Hartmann U, Manner N, Huijsmans J, Gossner L, Rabenstein T, Vieth M, Stolte M, Ell C. Long-term efficacy and safety of endoscopic resection for patients with mucosal adenocarcinoma of the esophagus. Gastroenterology. 2014 Mar;146(3):652-660.e1. doi: 10.1053/j.gastro.2013.11.006. Epub 2013 Nov 20. PMID 24269290
- [Background] Phoa KN, Pouw RE, Bisschops R, Pech O, Ragunath K, Weusten BL, Schumacher B, Rembacken B, Meining A, Messmann H, Schoon EJ, Gossner L, Mannath J, Seldenrijk CA, Visser M, Lerut T, Seewald S, ten Kate FJ, Ell C, Neuhaus H, Bergman JJ. Multimodality endoscopic eradication for neoplastic Barrett oesophagus: results of an European multicentre study (EURO-II). Gut. 2016 Apr;65(4):555-62. doi: 10.1136/gutjnl-2015-309298. Epub 2015 Mar 2. PMID 25731874
- [Background] Spechler SJ, Souza RF. Barrett's esophagus. N Engl J Med. 2014 Aug 28;371(9):836-45. doi: 10.1056/NEJMra1314704. No abstract available. PMID 25162890